CLINICAL TRIAL: NCT05834868
Title: A Phase 3, Randomized, Open-Label, Multicenter, Active-controlled Trial Comparing Efficacy and Safety of THDB0206 Injection With Insulin Lispro Injection Combined With Insulin Glargine Injection U-100 in Chinese Participants With Type 2 Diabetes
Brief Title: Efficacy and Safety of THDB0206 Compared to Insulin Lispro Injection in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THDB0206L02
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDB0206 Injection (Experimental)
  Interventions: Drug: THDB0206 Injection
- Insulin Lispro Injection (Active Comparator)
  Interventions: Drug: Insulin Lispro Injection

INTERVENTIONS:
Drug: THDB0206 Injection — Drug: THDB0206 Injection Injected subcutaneously three times a day. Dose was individually adjusted.
  Arms: THDB0206 Injection
Drug: Insulin Lispro Injection — Drug:Insulin Lispro Injection Injected subcutaneously three times a day. Dose was individually adjusted.
  Arms: Insulin Lispro Injection

SUMMARY:
This is a 26-week randomized, open-label, multicenter, active-controlled parallel group trial. The purpose of this study is to compare efficacy and safety of THDB0206 injection with insulin lispro injection combined with insulin glargine injection U-100 in Chinese participants with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: 18.0 kg/m^2~35.0 kg/m^2 (both inclusive) at the time of screening.
* HbA1c: 7.0%~10.0% (both inclusive) at the time of screening.
* Diagnosed with T2DM for 6 months or longer at the time of screening based on the World Health Organization (WHO) classification.
* Treated with stable insulin regimen as follow for at least 3 months with or without oral antidiabetic drug:

  1. Basal insulin (neutral protamine Hagedorn [NPH] insulin, insulin glargine, insulin degludec, insulin detemir) in combination with at least 1 prandial injection of bolus insulin.
  2. Premixed insulin at least twice daily.

Exclusion Criteria:

* Have other types of diabetes other than T2DM.
* Have used Glucagon-Like Peptide 1 (GLP-1) receptor agonist within 3 months prior to screening.
* Have had 1 or more episodes of severe hypoglycemia within the 6 months prior to screening.
* Have had 1 or more episodes of acute diabetic complications (diabetic ketoacidosis, hyperglycemic hyperosmolar state, diabetic lactic acidosis, etc.) within the 6 months prior to screening.
* With concomitant conditions at screening that may affect the evaluation of the study, including cardiovascular and cerebrovascular diseases, respiratory diseases, gastrointestinal diseases, liver diseases, kidney diseases, nervous system diseases, psychiatric diseases, hematological diseases, immune system diseases, endocrine system diseases, pancreatic diseases, and/or malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment | Week 26

SECONDARY OUTCOMES:
Change From Baseline in 1-hour Postprandial Glucose (PPG) Excursion at Week 26 | Week 26
Change From Baseline in 2-hour Postprandial Glucose (PPG) Excursion at Week 26 | Week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China